CLINICAL TRIAL: NCT03250481
Title: Responsiveness Index Versus the RASS Based Method for Adjusting Sedation in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Ville Pettilä, Professor, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HelsinkiUCHFin
Record Dates: First submitted 2017-08-08; First posted 2017-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Critical Illness
Keywords: Sedation, Responsiveness Index, Electromyogram
MeSH Terms: conditions — Critical Illness | interventions — Propofol; Oxycodone

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Sedation guidance with RASS-group (Active Comparator): Sedation is guided with RASS. Targeted sedation level is RASS -3 - 0. Propofol: an initial rate of 2.4 mg/kg/h for one hour. Thereafter, the infusion rate of propofol is 0.8-4 mg/kg/h to reach or maintain the target RASS score. Propofol bolus of 20-40 mg is allowed. Oxycodone as 3-6 mg boluses for pain management. Other opiates are not allowed. Midazolam may given if the maximum dose of propofol is reached and pain management by oxycodone restricted achievement of the target sedation level. Midazolam will supply intravenously in boluses of 1-2 mg (based on the weight of the patient), starting at 3 boluses/h for the first hour. Dexmedetomidine and other sedatives are not allowed.
  Interventions: Drug: Propofol
- 'Sedation guidance with RI (Experimental): Sedation is guided with RI. Targeted sedation level is RI 40-80. Propofol: an initial rate of 2.4 mg/kg/h for one hour. Thereafter, the infusion rate of propofol is 0.8-4 mg/kg/h to reach or maintain the target RI score. Propofol bolus of 20-40 mg is allowed. Oxycodone as 3-6 mg boluses for pain management. Other opiates are not allowed. Midazolam may given if the maximum dose of propofol is reached and pain management by oxycodone restricted achievement of the target sedation level. Midazolam will supply intravenously in boluses of 1-2 mg (based on the weight of the patient), starting at 3 boluses/h for the first hour. Dexmedetomidine and other sedatives are not allowed.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Sedation targeted to RASS -3-0 or RI 20-40
  Other Names: Oxycodone; Midazolame

SUMMARY:
Systematic evaluation of pain, agitation and delirium in ICU-patients is recommended and deep sedation should be avoided. Sedation is still monitored with clinical assessments, like RASS. The Responsiveness Index (RI) is a recently described method for ICU sedation monitoring. It is based on processed frontal EMG and reflects the interaction between a patient's conscious state and the intensity and frequency of stimulations during treatment. RI has not been randomly compared to RASS to titrate sedation to target at a clinically adequate sedation state. In this open randomized controlled pilot study of 32 critically ill, mechanically ventilated adult patients, investigators will evaluate the feasibility, safety and efficacy of RI based sedation compared to standard RASS based titration of sedation. Investigators hypothesize first that RI controlled sedation will be safe and, second that RI controlled sedation will associate with increased number of ventilator free days alive in 30 days without excess adverse events.

DETAILED DESCRIPTION:
Sedation of intensive care patients is needed for patient's safety but deep sedation is associated with adverse outcomes. Frontal electromyogram based Responsiveness Index (RI) aims to quantify patient's arousal. RI monitoring together with staff education may have potential to improve sedation quality. Investigators will evaluate the safety of RI based sedation versus standard care using Richmond Agitation-Sedation Scale (RASS) for sedation.

Methods: randomized study, critically ill adult patients with mechanical ventilation and administration of sedation to either RI- or RASS-guided sedation. Propofol (and midazolam combined with if needed) as a hypnotic drug and oxycodone as an analgesic drug. Investigators will follow standardized sedation protocol in both groups to achieve the predetermined target sedation level: either RI 40-80 (RI-group) or RASS -3-0 (RASS group). RI measurement is continuous in both groups, but blinded in the RASS group. Accordingly, RI group is blinded to RASS assessments. State Entropy (SE) will register in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care patients
* Need of mechanical ventilation and sedation

Exclusion Criteria:

* contraindication to propofol or oxycodone
* hypoxic or traumatic brain injury
* intracranial hemorrhage
* status epilepticus
* drug overdose as admission diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with sedation or sedation monitoring related predetermined adverse events | Up to 96 hours (starting when RI-monitoring begins)
  Predetermined adverse events hypotension, hypertension, tachycardia, tachypnea, anxiety, unintended catheter removal, gas exchange deficiency, skin irritation caused by electrodes, hemodynamic instability

SECONDARY OUTCOMES:
Increased ventilator free days | 30 days
  Time alive without mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Wennervirta, MD, PhD, Principal Investigator — University of Helsinki and Helsinki University Hospital, PO Box 340, 00029 Helsinki, Finland
Locations (1):
- HelsinkiUCH, Helsinki, Finland